CLINICAL TRIAL: NCT03257514
Title: Assessing The Effect of Alpha Lipoic Acid on Uterine Scar Healing After Cesarean Section by Using Saline Contrast Sonohysterography
Brief Title: Effect of Alpha Lipoic Acid on Uterine Scar Healing After Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: maternity hospital ASU
Record Dates: First submitted 2017-07-30; First posted 2017-08-22 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Cesarean Section; Dehiscence; Cesarean Scar Niche
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alpha lipoic acid (Active Comparator): 51 women will receive alpha lipoic acid drug (thiotacid film coated tablets 600 mg) for 6 weeks after cesarean section then uterine scar healing will be assessed by saline sonohysterography (by placing catheter in the cervical os helping to administering saline into uterine cavity then using the transvaginal ultrasound to view the uterus in the longitudinal view)
  Interventions: Drug: alpha lipoic acid drug (thioctic acid acid)
- placebo (Placebo Comparator): 51 women will receive a placebo drug for 6 weeks after cesarean section then uterine scar healing will be assessed by saline sonohysterography(by placing catheter in the cervical os helping to administering saline into uterine cavity then using the transvaginal ultrasound to view the uterus in the longitudinal view)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: alpha lipoic acid drug (thioctic acid acid) — Alpha lipoic acid has anti-inflammatory, antioxidant effects and plays a role in wound healing process.
  Arms: alpha lipoic acid
Drug: Placebo Oral Tablet — placebo oral drug have the same shape of thiotacid tablet
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of alpha lipoic acid on uterine scar healing after cesarean section by using saline contrast sonohysterography

DETAILED DESCRIPTION:
This is a triple blind randomized placebo controlled prospective clinical trial that will be conducted in Ain Shams University Maternity Hospital.

in which a consecutive series of participant attending emergency room 102 women undergoing cesarean section for the first time will be randomized into two groups.

Group A (Study group): 51 women will receive alpha lipoic acid drug ( 600 mg twice daily) for 6 weeks after cesarean section and saline sonohysterography will be done after that.

Group B (Control group): 51 women will receive a placebo drug twice daily for 6 weeks after cesarean section and saline sonohysterography will be done after that.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (gestational age between 37-41 weeks).
* Women undergoing cesarean section for the first time.
* Normal vaginal ultrasound examination and exclusion of any pelvic abnormality.
* Uncomplicated cesarean section.
* Lower uterine segment cesarean sections while the women not in labor.

Exclusion Criteria:

* Women with complications during or after cesarean section as intrapartum or postpartum hemorrhage, puerperal sepsis, septic wound
* Women with medical diseases that can affect the healing as diabetes mellitus, anemia, chronic renal disease or hepatic disease or coagulopathy or receiving medications affect wound healing as corticosteroids or anticoagulant.
* Women who will use intrauterine device as a contraceptive method
* Women with uterine abnormality as cervical stenosis or fibroid uterus
* Women with pelvic infection at the time of saline sonohysterography

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
presence of scar niche | six weeks after CS
  triangular shaped anechoic area at the site of incision
The healing ratio | six weeks after CS
  the thickness of residual myometrium covering the defect divided by the sum of the thickness of residual myometrium cover the defect and the height of wedge shaped defect

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Abbassia, Egypt